CLINICAL TRIAL: NCT01158924
Title: A Phase I/IIa, Multicenter, Open-label, Clinical Trial to Evaluate the Safety, Tolerability and Preliminary Effectiveness of Single Administration Intradiscal rhGDF-5 for the Treatment of Early Stage Lumbar Disc Degeneration
Brief Title: A Clinical Trial to Evaluate the Safety, Tolerability and Preliminary Effectiveness of Single Administration Intradiscal rhGDF-5 for the Treatment of Early Stage Lumbar Disc Degeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DePuy Spine (Industry)
Collaborators: Janssen-Cilag Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 09-Intradiscal rhGDF-5-02
Record Dates: First submitted 2010-07-01; First posted 2010-07-08 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Early Lumbar Disc Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intradiscal rhGDF-5 (Experimental): The API is recombinant human growth and differentiation factor-5 (rhGDF-5), a recombinant version of human GDF-5. GDF-5 is a member of the transforming growth factor-b (TGF-b) superfamily and the bone morphogenetic protein (BMP) subfamily, and is known to influence the growth and differentiation of various tissues, including the intervertebral disc. In vitro experiments have shown that rhGDF-5 can stimulate gene expression and synthesis of the extracellular matrix proteins type II collagen and aggrecan. In vivo experiments in rabbit models of disc degeneration have shown that intradiscal injections of rhGDF-5 can stimulate an increase in disc height and hydration.
  Interventions: Drug: Intradiscal rhGDF-5

INTERVENTIONS:
Drug: Intradiscal rhGDF-5 — The API is recombinant human growth and differentiation factor-5 (rhGDF-5), a recombinant version of human GDF-5. GDF-5 is a member of the transforming growth factor-b (TGF-b) superfamily and the bone morphogenetic protein (BMP) subfamily, and is known to influence the growth and differentiation of various tissues, including the intervertebral disc. In vitro experiments have shown that rhGDF-5 can stimulate gene expression and synthesis of the extracellular matrix proteins type II collagen and aggrecan. In vivo experiments in rabbit models of disc degeneration have shown that intradiscal injections of rhGDF-5 can stimulate an increase in disc height and hydration.

SUMMARY:
Study to show the safety, tolerability and preliminary effectiveness of Intradiscal rhGDF-5 in subjects with early lumbar disc degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent low back pain with at least 3 months of non-surgical therapy at one or two suspected symptomatic lumbar levels (L3/L4 to L5/S1)

   a. The recruiting physician will use their standard clinical and radiological practice to determine the one/two disc level(s) be treated, i.e., but not limited to a combination of MRI, CT and/or Technetium bone scans, functional x-rays, input from a spinal injection program (targeting facet joints and/or epidural space) and discography (a discogram performed within 12 months of the anticipated study treatment date is acceptable, as long as the subject has not had an accident or re-injury).
2. Oswestry Disability Index (ODI) for low back pain of 30 or greater
3. Low Back Pain score greater than or equal to 4 cm as measured by Visual Analog Scale (VAS) at Visit 1 Baseline
4. Male or Female 18 years of age or older

Exclusion Criteria:

1. Persons unable to have an MRI
2. Abnormal neurological exam at baseline (e.g., chronic radiculopathy)
3. Persons with neurological or radiographic evidence of active radicular pain due to anatomical compression such as stenosis or disc herniation (persons with somatic referred pain are allowed)
4. Suspected symptomatic facet joints and/or severe facet joint degeneration at the index level(s) or adjacent segments
5. Suspected symptomatic sacro-iliac joint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Hunter Clinical Research, Broadmeadow, New South Wales
  - St. George Private Hospital, Kogarah, New South Wales
  - BrizBain & Spine, The Wesley Hospital, Auchenflower, Queensland

RESULTS

PARTICIPANT FLOW:
Groups:
- Intradiscal rhGDF-5 (1.0mg); Intradiscal rhGDF-5 (2.0mg): The API is recombinant human growth and differentiation factor-5 (rhGDF-5), a recombinant version of human GDF-5. GDF-5 is a member of the transforming growth factor-b (TGF-b) superfamily and the bone morphogenetic protein (BMP) subfamily, and is known to influence the growth and differentiation of various tissues, including the intervertebral disc.
Period: Overall Study
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Intradiscal rhGDF-5 (2.0mg)
Started | 14 | 26
Completed | 13 | 23
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Intradiscal rhGDF-5 (2.0mg) | Total
Number analyzed (Participants) | 14 | 26 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (10.85) | 48.3 (10.37) | 46.9 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 6 | 15 | 21
Region of Enrollment [Number; unit: participants]
  Australia | 14 | 26 | 40

OUTCOME MEASURES:

1. Primary Outcome: Neurological Assessment for Motor Function and Reflexes/Sensory
Description: Neurological Assessment for Motor Function and Reflexes/Sensory- Number of patients with Clinically Significant Abnormal results at 12 months.
  For Motor Function, Clinically Significant Abnormal results are determined by the surgeon investigator and are further classified by grade: 0= No Movement, 1= Flicker/trace of contraction, 2=Active movement when gravity removed, 3= Active movement against gravity, 4= Active Movement against gravity and resistance.
  For Reflexes/Sensory, Clinically Significant Abnormal results are determined by the surgeon investigator and are based on exams of the Knee, Ankle, L3-L5 Dermatone, and S1 Dermatome. Tension signs are evaluated with a straight leg raise to determine at which point, if any, sciatic pain occurs.
Time Frame: 12 months
Population: Safety Population
  The Neurological Assessment at 12 months was only conducted on 13 subjects from the 1.0mg group (out of 14 total subjects) and 25 subjects from the 2.0 mg group (out of 26 total).
Measure: Number; unit: participants
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Intradiscal rhGDF-5 (2.0mg)
Number analyzed (Participants) | 13 | 25
participants | 0 | 2

2. Secondary Outcome: Change in Function Assessed by Oswestry Disability Index Change at 12 Months From Baseline
Description: The Oswestry Disability Index (ODI) is a 10-category (Pain Intensity, Personal Care, Lifting, Walking, Sitting, Standing, Sleeping, Sex Life, Social Life, Traveling) disability measurement scale with a graded response from 0 to 5, with 0 being the best score (no impairment) to 5 being the worst score (significant impairment). ODI score for a subject is calculated by adding the scores and converting the score to a 100 point scale.
Time Frame: 12 months
Population: FAS Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Intradiscal rhGDF-5 (2.0mg)
Number analyzed (Participants) | 14 | 26
units on a scale | -13.0 (14.63) | -18.1 (13.69)

3. Primary Outcome: Treatment Emergent Adverse Events- Relationship to Study Drug
Description: Number of patients with Treatment Emergent Adverse Events that were designated as related or possibly related to Study Drug.
Time Frame: Through a 12 month period and annual telephone contact at 24 and 36 months for subject health status follow-up.
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Intradiscal rhGDF-5 (2.0mg)
Number analyzed (Participants) | 14 | 26
participants | 2 | 1

4. Secondary Outcome: Change in Pain Visual Analog Scale (VAS) at 12 Months From Baseline.
Description: The Visual Analog Scale (VAS) pain score asks the subject to place a vertical mark on a horizontal line (that is approximately 10 cm long) with 'No Pain' (score of 0 = 0 cm) listed on the left and 'Very severe pain' (score of 10=10cm) labeled on the right. The subject is instructed to indicate the amount of pain they feel in their back.
Time Frame: 12 months
Population: FAS Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Intradiscal rhGDF-5 (2.0mg)
Number analyzed (Participants) | 14 | 26
units on a scale | -2.66 (3.448) | -3.80 (2.651)

5. Secondary Outcome: Change in Physical Component Summary of Quality of Life Measure Assessed by Short-Form 36 at 12 Months From Baseline.
Description: The 36-item Short Form Health Survey (SF-36) is a patient reported outcome survey that evaluates functional health and well-being. The survey is converted into two summary measures (the Physical Component - PCS and Mental Component- MCS) that are scored from 0 to 100 (where 100 indicates the highest level of health).
Time Frame: 12 Months
Population: FAS Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Intradiscal rhGDF-5 (2.0mg)
Number analyzed (Participants) | 14 | 26
units on a scale | 11.18 (13.206) | 10.00 (9.897)

ADVERSE EVENTS:
Time Frame: Adverse events were collected through a 12 month period and annual telephone contact at 24 months and 36 months
Arm/Group | Intradiscal rhGDF-5 (1.0mg) | Intradiscal rhGDF-5 (2.0mg)
Serious Adverse Events (participants affected / at risk) | 1/14 | 4/26
Other Adverse Events (participants affected / at risk) | 12/14 | 18/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intradiscal rhGDF-5 (1.0mg) (N=14) | Intradiscal rhGDF-5 (2.0mg) (N=26)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Guillain-Barre Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intradiscal rhGDF-5 (1.0mg) (N=14) | Intradiscal rhGDF-5 (2.0mg) (N=26)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (7) | 12 (20)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Staphlococcal Infection (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
Migraine (Nervous system disorders) | 3 (5) | 1 (2)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subcutaneous Nodule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Oropharyngeal Spasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Seasonal Allergy (Immune system disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Investigators may freely present or publish results of the Clinical Investigation in a manner which fairly sets forth the conclusions reached by the Clinical Investigators, but only after the Sponsor has been given the opportunity of reviewing the proposed presentation or publication at least 60 days prior to the intended submission, presentation, or publication date.